CLINICAL TRIAL: NCT05732246
Title: Effect of First Rib Mobilization With Balloon Breathing Exercises in Non Specific Chronic Neck Pain: A Randomized Control Trial
Brief Title: Effect of First Rib Mobilization With Balloon Breathing Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ferozanawaz15
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment group (No Intervention): Hot pack and TENS at neck for 10minutes. Therapeutic ultrasound for 5 minutes Soft tissue techniques (gliding and kneading) was applied at a slow speed for 5 minutes over the neck muscles.
  Gentle stretching and strengthening exercises
- First rib mobilization with balloon breathing exercises group (Experimental): Patient was in supine position, placing the soles of his feet against the wall so that the ankle, knee, and thigh joints are at a 90-degree angle. The subject placed a 3-4-inch ball between his/her knees, which he/she has to maintain through the pressure of the internal thigh muscles during the whole training period and puts his/her back on the bed. Holds the right hand above the head and the left hand with the balloon. Meanwhile examiner palpated 1st rib with head in left side flexion. Patient was then asked to inhale through the nose in three-four seconds and then exhales slowly into the balloon. Then, holding the first rib in place, the patient was asked to inhale and exhale deeply again. The examiner continued applying pressure to hold the first rib in a position of relative depression during inhalation, and further depress the first rib as able during exhalation.
  Interventions: Other: First rib mobilization with balloon breathing exercises

INTERVENTIONS:
Other: First rib mobilization with balloon breathing exercises — Patient was in the supine position, placing the soles of his feet against the wall so that the ankle, knee, and thigh joints are at a 90-degree angle. The subject placed a 3-4-inch ball between his/her knees, which he/she has to maintain through the pressure of the internal thigh muscles during the whole training period and puts his/her back on the bed. Holds the right hand above the head and the left hand with the balloon. Meanwhile examiner would palpate 1st rib with head in left side flexion. Patient was then asked to inhale through the nose in three-four seconds and then exhales slowly into the balloon. Then, holding the first rib in place, the patient was asked to inhale and exhale deeply again. The examiner continued applying pressure to hold the first rib in a position of relative depression during inhalation, and further depressed the first rib as able during exhalation.
  Arms: First rib mobilization with balloon breathing exercises group

SUMMARY:
As Non specific chronic neck pain is effecting quality of life in many ways, there are many studies evaluating the methods to treat that problem. This study aims to determine Effect of first rib mobilization with balloon breathing exercises in non specific chronic neck pain. Patients would be divided into two groups and both received conventional treatment. Group A got conventional treatment only but Group B got 1st rib mobilization with balloon breathing exercises in addition.

DETAILED DESCRIPTION:
Nonspecific chronic neck pain (NSCNP) is defined as neck pain persisting for longer than 12 weeks or after the healing period or recurring neck pain that intermittently affects an individual over a long time. Due to current life style, 22 to 70% of the population is expected to feel neck pain somewhere in their lives.

People with non-specific chronic neck pain (NSCNP) present with local hyperalgesia, impaired conditioned pain modulation, low quality of life, and psychological disruptions (fear of movement, depressive symptoms, pain catastrophizing) A systematic review and meta-analysis on Respiratory dysfunction in patients with chronic neck pain reports that, patients with Chronic Neck Pain have reduced respiratory muscle strength and pulmonary function compared with asymptomatic individuals, and this difference could be clinically meaningful.

As previous studies provides evidence about effect of MWM on non specific chronic neck pain and also states relation of breathing dysfunction in NSCNP so we aim to determine effect of first rib mobilization with balloon breathing exercise in addition to conventional treatment in non specific chronic neck pain.

Patients would be divided into two groups and both received conventional treatment. Group A got conventional treatment only but Group B got 1st rib mobilization with balloon breathing exercises in addition.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18-45 years
* Gender: Male, Female
* Patients with non-specific chronic neck pain referred by physician or orthopedic surgeon
* Computer users, mobile users and those with routine of prolonged sitting

Exclusion Criteria:

* Any H/o neurological or vestibular disorders.
* Any H/o Cervical Trauma or surgery
* Any history of Physiotherapy treatment for the cervical region within the previous three months
* cardiac or respiratory insufficiency
* Pregnancy
* Neoplasm

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (change is being assessed) | Change from Baseline measures at 8 weeks
  Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. 0-4points (0-8%) no disability, 5-14points ( 10 - 28%) mild disability, 15-24points (30-48% ) moderate disability, 25-34points (50- 64%) severe disability, 35-50points (70-100%) complete disability
Numeric Pain Rating Scale (change is being assessed) | Change from Baseline measures at 8 weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"
Single Breath Count (change is being assessed) | Change from Baseline measures at 8 weeks
  Participants will be requested to count out loud after maximal inspiration. The ability to reach a count of 50 is considered as normal respiratory function
Chest Wall Expansion (change is being assessed) | Change from Baseline measures at 8 weeks
  Take an inches tape and encircle chest around the level of nipple. Take measurements at the end of deep inspiration and expiration.
  Normally, a 2-5" of chest expansion can be observed

CONTACTS AND LOCATIONS:
Overall Officials: Feroza Nawaz, MSOMPT, Principal Investigator — University of Lahore
Locations (1):
- Sehat Medical Complex, Lahore, Lahore, Punjab Province, Pakistan